CLINICAL TRIAL: NCT06669975
Title: A Phase 1/2, Open-label Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of AP402 in HER2-Positive Patients With Locally or Advanced Solid Tumors
Brief Title: A Study of AP402 in HER2-Positive Patients With Locally or Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AP Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP402-101
Record Dates: First submitted 2024-10-10; First posted 2024-11-01 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor
Keywords: HER2-positive; local solid tumors; advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose escalation) (Experimental)
  Interventions: Drug: AP402 (Part 1 Dose esclation)
- Part 2 (Dose Expansion) (Experimental)
  Interventions: Drug: AP402 (Part 2 Dose Expansion)

INTERVENTIONS:
Drug: AP402 (Part 1 Dose esclation) — Dose escalation will consist of 7 cohorts where an Intraveous infusion of AP402 will be administered once every 2 weeks to determine the maximum tolerated dose (MTD) (ie, the highest safe dose administered to patients) and the recommended phase 2 dose (RP2D) of AP402.
  Arms: Part 1 (Dose escalation)
Drug: AP402 (Part 2 Dose Expansion) — After the MTD and/or RP2D are determined by the SRC, additional patients will be enrolled in Phase 2 dose expansion and will be treated with AP402 at that dose.
  Arms: Part 2 (Dose Expansion)

SUMMARY:
This is a Phase 1/2, multi-regional, multi-center, open-label, first-in-human (FIH), dose-escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary clinical activity of AP402 in HER2-positive patients with locally or advanced solid tumors.

DETAILED DESCRIPTION:
The study will consist of 2 parts:

* Part 1 (Dose Escalation): Dose escalation will consist of 7 cohorts where an IV infusion of AP402 will be administered once every 2 weeks to determine the maximum tolerated dose (MTD) (ie, the highest safe dose administered to patients) and the recommended phase 2 dose (RP2D) of AP402. For dose-escalation, an accelerated dose titration design will be utilized for the first 2 dose cohorts, followed by a standard 3+3 dose titration design for the remaining 5 cohorts. Up to 42 patients will be enrolled in Part 1.
* Part 2 (Dose Expansion): After the MTD and/or RP2D are determined by the Safety Review Committee (SRC) (see Section 6.5), additional patients will be enrolled in Part 2 and will be treated with AP402 at that dose once every 2 weeks. Part 2 will be based on the Simon's two-stage optimal design (Simon, 1989) and is expected to enroll approximately 43 patients in 1 or 2 selected tumor types.

Administration of the IP will continue for 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, intolerable toxicity, withdrawal of consent, study completion, death or other reasons leading to treatment discontinuation, whichever comes first

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically proven locally unresectable advanced or metastatic HER2-postive solid tumors which no standard therapy suitable.
2. Adult patients aged ≥ 18 years at the time of signing informed consent form (ICF).
3. Written informed consent by the patients or the patient's legally authorized representative prior to Screening.
4. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at study enrollment and an estimated life expectancy of at least 3 months.
5. Disease must have at least 1 measurable (long diameter ≥ 1cm) lesion by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Tumor lesions situated in a previously irradiated area are not considered assessable unless there has been demonstrated progression in the lesion. Imaging tests outside the screening period are valid if performed not more than 2 weeks before consent signature and otherwise fulfil protocol criteria.
6. Patients with adequate organ function defined by the following:

   1. Absolute neutrophil count ≥ 1.5 × 109 /L.
   2. Platelet count ≥ 100 × 109 /L.
   3. Hemoglobin ≥ 9 g/dL.
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN or < 5 × ULN if hepatic metastases present.
   5. Serum total bilirubin ≤ 1.5 × ULN (or < 3 × ULN for patients with Gilbert's syndrome).
   6. Alkaline phosphatase ≤ 2.5 × ULN or < 5 × ULN if bone metastases present.
   7. Prothrombin time ≤ 1.5 × ULN.
   8. International normalized ratio (INR) ≤ 2.0 or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Exception: INR 2 to ≤ 3 is acceptable for patients on a stable dose of anticoagulants.
   9. Estimated creatinine clearance > 45 mL/min according to the Cockcroft Gault formula.
   10. Albumin ≥ 28 g/L NOTE: Patients must not have required blood transfusions or growth factor support ≤ 14 days before sample collection at Screening.
7. Females must not be pregnant or lactating, and must use acceptable, highly effective double contraception from Screening until 90 days after study completion, including the Follow-up period. Effective forms of contraception are defined in Section 7.3.2. Females with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study. Women not of childbearing potential must be postmenopausal for ≥12 months (postmenopausal status is to be confirmed through testing of FSH levels ≥ 40 IU/L at Screening for amenorrhoeic female patients).
8. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), or if engaged in sexual relations with a WOCBP, either his partner must be surgically sterile (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or an acceptable, highly effective contraceptive method (see Section 7.3.2) must be used from Screening until study completion, including the Follow-up period. Males with same-sex partners (abstinence from penile-vaginal intercourse) or are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle. Males must not donate sperm from the first dose of IP until at least 90 days after the last dose of IP.

Exclusion Criteria:

1. Patients who have received concurrent antitumor treatment or investigational products within 28 days or 5 half-lives before the start of IP, whichever comes earlier. The antitumor treatments include chemotherapy, radiotherapy (with the exception of palliative bone directed radiotherapy), immunotherapy, targeted therapy, hormonal therapy, or cytokine therapy except for erythropoietin.
2. Patients who had received CD137-targeted therapeutics within 28 days or 5 half-lives before the start of IP, whichever comes earlier.
3. Patients who had major surgery within 28 days before the start of IP (excluding prior diagnostic biopsy).
4. Patients who had continuance of toxicities due to prior antitumor agents that have not resolved to Grade ≤ 1 per NCI CTCAE version 5.0, except alopecia, and< Grade 2 sensory neuropathy.
5. Patients with a history of immune mediated AE of any grade that resulted in discontinuation of prior immunotherapy.
6. Patients with previous malignant disease other than the target malignancy to be investigated in this study within the last 2 years with the exception of resected basal or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix or breast.
7. Patients with active leptomeningeal disease or uncontrolled, untreated brain metastasis. Patients with a history of treated and, at the time of Screening, stable central nervous system (CNS) metastases are eligible, provided they meet all the following:

   1. Brain imaging at Screening shows no evidence of interim progression, patient is clinically stable for at least 2 weeks and without evidence of new brain metastases.
   2. Measurable disease outside the CNS.
   3. No ongoing requirement for corticosteroids as therapy for CNS disease; off steroids 2 weeks before the first dose of AP402; anticonvulsants at a stable dose are allowed.
8. Patients who received any organ transplantation including allogeneic stem cell transplantation.
9. Patients with significant acute or chronic infections including, among others:

   1. Infection requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days before first dose of AP402.
   2. Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
   3. Note: An HIV serology test (including antigen and/or antibodies) will be conducted at baseline for the patients with unknown HIV status and patients with positive HIV test will be excluded.
   4. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV deoxyribonucleic acid (DNA) > 500 IU/mL (or > 2500 copies/mL) at Screening.
   5. NOTE: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL or < 2500 copies/mL) can be enrolled. Patients with detectable HBsAg or detectable HBV DNA should be managed per treatment guidelines. Patients receiving antivirals at Screening should have been treated for > 2 weeks before the first dose of AP402.
   6. Patients with active hepatitis C.
   7. NOTE: Patients with a negative hepatitis C virus (HCV) antibody test at Screening or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at Screening are eligible. The HCV RNA test will be performed only for patients testing positive for HCV antibody. Patients receiving antivirals at Screening should have been treated for > 2 weeks before the first dose of AP402.
10. Patients with active or history of any autoimmune disease that may relapse (patients with diabetes Type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible) or immunodeficiencies. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of AP402.
11. Patients with known severe hypersensitivity reactions to monoclonal antibodies.
12. Patients with pregnancy or lactation period. Note: a negative pregnancy test is required for WOCBP.
13. Patients with known alcohol or drug abuse.
14. Patients with clinically significant (ie, active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to the first dose of AP402), myocardial infarction (< 6 months prior to the first dose of AP402), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication, or baseline QTcF interval > 480 msec.
15. Patients with a left ventricular ejection fraction (LVEF) lower than 55% at Screening.
16. Patients with any psychiatric condition that would prohibit the understanding or rendering of informed consent.
17. Patients with live (or live attenuated) vaccination within 28 days of the first dose of AP402 and during the study period.
18. NOTE: COVID-19 vaccinations are permitted while a patient is on the study.
19. Patients with all other significant diseases, in the opinion of the Investigator, might impair the patient's tolerance of the IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Estimate of Maximum tolerated dose (MTD) | Baseline to 90 days after the last dose
  This will be based on dose limiting toxicities (DLT) observed during the DLT evaluation period.
Number of participants with Adverse events (AEs) and Serious Adverse events (SAE) as assessed by CTCAE V5 | Baseline to 90 days after the last dose
To evaluate R2PD based on PK parameters- Cmax (Maximum plasma concentration) | Baseline to 90 days after the last dose
To evaluate R2PD based on PK parameters- Tmax (time for maximum concentration) | Baseline to 90 days after the last dose
To evaluate R2PD based on PK parameters- AUC (Area under curve) | Baseline to 90 days after the last dose
To evaluate R2PD based on PK parameters- T1/2 (terminal half-life) | Baseline to 90 days after the last dose

SECONDARY OUTCOMES:
To evaluate objective response rate (ORR) | Baseline to 30 days after the last dose
  The proportion of patients whose best overall response (BOR) is either confirmed complete responses (CR) or confirmed partial responses (PR).
Number of patients with disease Control Rate (DCR) | Baseline to 90 days after the last dose
  The proportion of patients whose best overall response of confirmed CR, confirmed PR, or (confirmed) stable disease (SD) that was assessed at least 4 weeks (28 days) following the initiation of AP402
Number of patients with changes in duration of objective response (DOOR) | Baseline to 30 days after the last dose
  The time from first documented objective response (confirmed CR or confirmed PR) until the earlier of disease progression or death from any cause, whichever occurs first.
Duration of disease control response (DODC): | Baseline to 30 days after the last dose
  The time from first documented disease control response (confirmed CR, confirmed PR, or confirmed SD) until the earlier of disease progression or death from any cause, whichever occurs first. This will only be applicable for patients who have a confirmed best overall response of CR, PR, or SD. Patients without the events (progressive disease or death) will be censored at the date of their last tumor assessment.
To assess progression-free survival (PFS): | Up to 48 months
  The time from start of study treatment to the earlier of either disease progression or death from any cause, whichever occurs first.
To assess overall Survival (OS) | Up to 48 months
  The time from start of study treatment to the date of death from any cause. Patients alive will be censored at the date of last known alive.
To assess time to Objective Response (TTOR): | Baseline to 30 days after the last dose
  The time from start of study treatment to the first documented objective response (confirmed CR or confirmed PR), whichever occurs first.
To assess time to disease control response (TTDC): | Baseline to 30 days after the last dose
  The time from start of study treatment to the first documented disease control response (confirmed CR, confirmed PR, or confirmed SD (at least 4 weeks (28 days) following the initiation of AP402)), whichever occurs first.
Serum concentration of AP402 | Baseline to 30 days after the last dose
To evaluate immunogenicity by the number and percentage of patients who develop ADA | Baseline to 30 days after the last dose
To evaluate immunogenicity by the number and percentage of patients who develop neutralizing antibodies (if applicable). | Baseline to 30 days after the last dose

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Macquarie University Clinical Trials Unit, Macquarie, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Linear Clinical Research, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No